CLINICAL TRIAL: NCT07165769
Title: Zanubrutinib, Obinutuzumab, and Lenalidomide (ZGR) in the Treatment of Newly Diagnosed Splenic B-cell Lymphoma With Prominent Nucleoli (SBLPN): A Prospective, Open-label, Single-arm Clinical Trial
Acronym: ZGR in SBLPN
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2025004
Record Dates: First submitted 2025-09-03; First posted 2025-09-10 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-09

CONDITIONS: Splenic B-cell Lymphoma/Leukaemia With Prominent Nucleoli，SBLPN
MeSH Terms: interventions — Neoadjuvant Therapy; Maintenance

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Induction therapy and maintenance therapy of BGR (Experimental): 1. Induction Therapy Induction Therapy consists of zanubrutinib plus lenalidomide: each cycle lasts 28 days, up to 6 cycles, followed by maintenance therapy.
  2. Maintenance Therapy Maintenance therapy consists of zanubrutinib plus lenalidomide: Lenalidomide is continued for 1 year. Zanubrutinib is continued for 2 years.
  Interventions: Drug: Induction Therapy; Drug: Maintenance Therapy

INTERVENTIONS:
Drug: Induction Therapy — All enrolled patients will receive the ZGR regimen (zanubrutinib, obinutuzumab, and lenalidomide) for induction therapy. Each cycle lasts 28 days, up to 6 cycles, followed by maintenance therapy. Patients experiencing disease progression during induction will discontinue the trial drugs but remain under survival follow-up.
  1. Zanubrutinib: 160 mg twice daily, administered orally continuously.
  2. Obinutuzumab: 1000 mg via intravenous infusion, administered on Days 1, 8, and 15 of Cycle 1 and subsequently on Day 1 of Cycles 2-6.
  3. Lenalidomide: 25 mg once daily, taken orally on Days 1-21 of each 28-day cycle until disease progression. Doses should be taken at approximately the same time daily.
Drug: Maintenance Therapy — Maintenance therapy consists of zanubrutinib plus lenalidomide:
  Lenalidomide is continued for 1 year. Zanubrutinib is continued for 2 years. Treatment continues until disease progression, intolerability, or completion of 2 years. For patients who do not achieve complete remission (CR), therapy may continue until progression or intolerability.
  1. Zanubrutinib: 160 mg twice daily, administered orally continuously.
  2. Lenalidomide: 10 mg once daily, taken orally on Days 1-21, followed by a 7-day rest period, constituting a 28-day cycle.

SUMMARY:
:The aim of this study was to analyze the safety and efficacy of Zanubrutinib, Obinutuzumab, and Lenalidomide (ZGR) in the Treatment of Newly Diagnosed Splenic B-cell Lymphoma with Prominent Nucleoli (SBLPN).

The main questions it aims to explore the Preliminary Efficacy of the Zanubrutinib, Obinutuzumab, and Lenalidomide (ZGR) Regimen in the Treatment of Newly Diagnosed SBLPN Patients.

To explore the safety of zanubrutinib, obinutuzumab combined with lenalidomide (ZGR) in the treatment of newly diagnosed SBLPN patients.

DETAILED DESCRIPTION:
There is no consensus on optimal first-line therapy for splenic B-cell lymphoproliferative neoplasms (SBLPN). Existing regimens like cladribine/bendamustine plus rituximab face toxicity and resistance. Targeting Bruton's tyrosine kinase (BTK), the novel BTK inhibitor zanubrutinib (highly selective, low toxicity) combined with obinutuzumab (enhanced antibody-dependent cytotoxicity) and lenalidomide (immunomodulation) shows promise. This single-arm trial evaluates the ZGR regimen (zanubrutinib, obinutuzumab, lenalidomide) for untreated SBLPN, including 6-cycle induction and maintenance therapy (zanubrutinib-lenalidomide), aiming to enhance efficacy, survival, and tolerability, offering a novel approach for this rare disease.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 80 years, male or female
* Histologically or cytologically confirmed SBLPN requiring active treatment;
* No prior systemic therapy for SBLPN received;
* ECOG performance status of 0-2;
* Anticipated life expectancy ≥6 months;
* Laboratory parameters (hematologic and biochemical) meeting the following criteria:
* a. Absolute neutrophil count (ANC) ≥1.0 × 10⁹/L, platelet count ≥50 × 10⁹/L;
* b. Total bilirubin (TBIL) ≤2.0 × upper limit of normal (ULN);
* c. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 × ULN;
* d. Creatinine clearance ≥50 mL/min (calculated via Cockcroft-Gault formula or direct measurement).
* Men and women of childbearing potential must agree to use medically approved contraception throughout the study and for 4 weeks after treatment discontinuation;
* Participants must voluntarily enroll in the study and provide written informed consent.

Exclusion Criteria:

* History of central nervous system (CNS) disorders (including CNS lymphoma) diagnosed within 1 year prior to enrollment.
* Other primary malignancies within the past 3 years (excluding non-melanoma skin cancer, curatively treated localized prostate cancer, cervical carcinoma in situ, or squamous intraepithelial lesions on PAP smear).
* Exposure to any investigational drugs, antimicrobial agents, or participation in other interventional clinical trials within 4 weeks prior to enrollment.
* Major surgery (excluding lymph node biopsy) within 14 days before enrollment or anticipated requirement for major surgery during the study.
* Prior use of investigational agents targeting SBLPN.
* Active immunodeficiency, autoimmune diseases, prolonged systemic corticosteroid therapy (>10 mg/day prednisone equivalent) within 7 days prior to enrollment, or any immunosuppressive therapy.
* Severe hepatic dysfunction (e.g., severe jaundice, hepatic encephalopathy, refractory ascites, hepatorenal syndrome), cachexia, multiorgan failure, or severe renal impairment.
* Clinically significant cardiovascular comorbidities:

New York Heart Association (NYHA) class III/IV heart failure; Myocardial infarction within 6 months prior to enrollment; Uncontrolled arrhythmias (including QTc interval ≥480 ms); Poorly controlled hypertension (systolic ≥150 mmHg/diastolic ≥100 mmHg despite antihypertensives); Unstable angina.

* Bleeding diathesis or coagulation disorders; thrombotic events within 3 months prior to enrollment.
* Hypersensitivity to active ingredients or excipients of the investigational drugs.
* Pregnancy, lactation, or women of childbearing potential unwilling/unable to use contraception.
* Other conditions deemed unsuitable for participation by the investigator (e.g., compromised protocol compliance or safety risks).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2025-09-04 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate，ORR | up to the end of 9 cycles of treatment(each cycle is 28 days)]
  defined as the proportion of patients with complete or partial response as assessed by response to induction therapy.

SECONDARY OUTCOMES:
complete response rate，CRR | Up to the end of 9 cycles of treatment(each cycle is 28 days)
progression-free survival，PFS | up to 5 years
  defined as the time from the start of treatment to disease progression or death due to any cause
duration of response，DOR | up to 5 years
  defined as the time from the first treatment response (including complete response and partial response) to the last assessment of response.
Overall survival，OS | Up to 5 years
  Defined as the time from enrollment to death for any cause.
Minimal Residual Disease，MRD | Up to the end of 2 years (each cycle is 28 days)
Adverse event rate | Up to the end of 2 years (each cycle is 28 days)

CONTACTS AND LOCATIONS:
Overall Officials: Shuhua Yi, Dr, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (1):
- Institute of Hematology and Blood Diseases Hospital ,Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No